CLINICAL TRIAL: NCT00626756
Title: LIGA Trial-Lithium Dilution Method in Guiding Fluid Therapy in Critically Ill Patients
Brief Title: Lithium Dilution Method in Guiding Fluid Therapy in Critically Ill Patients
Acronym: LIGA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: ASQA a.s. (Industry)
Responsible Party: Pavel Valek M.D., ASQA a.s.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: LigaStudy; LIGA2008
Record Dates: First submitted 2008-02-21; First posted 2008-02-29 (Estimated); Last update posted 2008-02-29 (Estimated); Status verified 2008-02

CONDITIONS: Critical Illness
Keywords: fluid; Lidco technology; guided therapy; fluid management guided by Lidco technology
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LI (Experimental): arm controled by LIDCO technology
  Interventions: Device: LiDCO technology
- CA (No Intervention): standard approach

INTERVENTIONS:
Device: LiDCO technology — non invasive monitoring of cardiac output
  Arms: LI

SUMMARY:
Hypothesis: Fluid management guided by LiDCO doesn´t increase cumulative fluid balance and shorten organ dysfunction compared to fluid management based on CVP and clinical judgment.

ELIGIBILITY:
Inclusion Criteria:

* Age
* Needs for fluid chalange
* Invasive ventilatory supportinvasive blood pressure monitoring
* Lidco monitoring
* Central venous catheter

Exclusion Criteria:

* DNR
* Need for CRRT
* Head injury

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2008-01; Primary Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
positive or negative fluid balance | one year

SECONDARY OUTCOMES:
effect of LiDCO monitoring on cumulative fluid balance | one year

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Cerny, MD, PhD, FCCM, Principal Investigator — University Hospital Hradec Kralove
Locations (1):
- ASQA a.s., Prague, Czechia

REFERENCES:
- [Background] Sinclair S, James S, Singer M. Intraoperative intravascular volume optimisation and length of hospital stay after repair of proximal femoral fracture: randomised controlled trial. BMJ. 1997 Oct 11;315(7113):909-12. doi: 10.1136/bmj.315.7113.909. PMID 9361539
- [Background] Wakeling HG, McFall MR, Jenkins CS, Woods WG, Miles WF, Barclay GR, Fleming SC. Intraoperative oesophageal Doppler guided fluid management shortens postoperative hospital stay after major bowel surgery. Br J Anaesth. 2005 Nov;95(5):634-42. doi: 10.1093/bja/aei223. Epub 2005 Sep 9. PMID 16155038
- [Background] Price J, Sear J, Venn R. Perioperative fluid volume optimization following proximal femoral fracture. Cochrane Database Syst Rev. 2002;(1):CD003004. doi: 10.1002/14651858.CD003004. PMID 11869649
- [Background] Price JD, Sear JW, Venn RM. Perioperative fluid volume optimization following proximal femoral fracture. Cochrane Database Syst Rev. 2004;(1):CD003004. doi: 10.1002/14651858.CD003004.pub2. PMID 14974001
- [Background] Conway DH, Mayall R, Abdul-Latif MS, Gilligan S, Tackaberry C. Randomised controlled trial investigating the influence of intravenous fluid titration using oesophageal Doppler monitoring during bowel surgery. Anaesthesia. 2002 Sep;57(9):845-9. doi: 10.1046/j.1365-2044.2002.02708.x. PMID 12190747